CLINICAL TRIAL: NCT05640700
Title: Assessing Personalized Vaginal Microbiome Contributions to HPV-driven Pre-malignant and Malignant Cervical Cancer
Brief Title: Vaginal Microbiome and HPV Pre-malignant and Cervical Dysplasia
Status: Recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ahinoam Lev-Sagie, Professor, Hadassah Medical Organization
Other Study IDs: HMO-812-21
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Human Papilloma Virus; Vaginal Flora Imbalance; Cancer Cervix Uterus; Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal for microbiome and molecular analysis, cytology and HPV PCR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Controls: Healthy women without HPV in their cervical and vaginal sample
- Women with HPV: Women with HPV, with or without cervical intraepithelial neoplasia or carcinoma

SUMMARY:
In this study, the investigators will prospectively collect, analyze and integrate information regarding vaginal microbiome composition and HPV presence in women with cervical pathologies (high-grade CIN and CC) and controls, to construct a large dataset from patients with pre-cancerous cervical lesions and healthy women, to evaluate the personalized contribution of the vaginal microbiome to the CIN-CC sequence.

DETAILED DESCRIPTION:
Infection with high-risk Human Papillomavirus (HPV) genotypes constitutes a well-recognized risk factor for cervical-carcinoma (CC). High-risk HPV features 10-15% persistence rate, consequently driving precancerous cervical-intraepithelial-neoplasia (CIN) and subsequent progression to CC. Multiple factors are believed to play permissive roles in the progression of CIN/CC , yet a molecular mechanism driving carcinogenesis across the CIN-CC continuum following persistent HPV infection remains elusive. The vaginal microbiome may play a role in the development of CIN-CC carcinogenesis, by modulation of host-immune-response and alteration of cervical microenvironment to become tumor-permissive. While suggested vaginal microbiome contributions include induction of altered epithelial cell adhesion and downregulation of DNA damage responses, no clear mechanism has been proven to date. The loss of Lactobacillus genus dominancy, and the switch to dysbiotic, high-diversity, high-pH, Bacterial Vaginosis (BV) is thought to play a key-role in HPV infection, persistence and carcinogenesis.

the investigators hypothesize that specific vaginal microorganisms may promote HPV persistence, chronic inflammation and progression through the CIN-CC sequence, and the elimination of harmful bacteria or supplementation of beneficial microbes, could possibly reverse HPV persistency and inhibit CIN-CC progression.

The current study consists of recruitment of a human cohort of healthy, CIN and CC patients including vaginal samples and comprehensive metadata collection. The investigators plan to conduct an in-depth characterization of vaginal microbiome to identify associations with HPV, CIN and CC.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-70
* Attended the clinic for a Pap smear or colposcopy

Exclusion Criteria:

* Patient does not approve sample collection
* Usage of antibiotics in the month prior to clinic visit
* Usage of any vaginal preparation or medication in the week prior to sample collection (anti-fungal, spermicides, lubricant etc.)
* Menstruation
* Pregnancy

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — people with cervix uterus
Study Population: 1) Individuals that underwent an HPV PCR cervical screening test and were found to be negative for HPV (healthy controls, n=45) 2) Women that were found to be positive for high risk-HPV but have no cervical dysplasia (n=30) 3) Women who are positive for high risk-HPV and exhibit cervical pathology, either high-CIN (CIN 2-3) or CC (n=15).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Characterization of the microbiome using molecular methods. | 1 year
  Comparison of microbiome profiles between those with HPV compared to controls without HPV.

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam Lev Sagie, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No